CLINICAL TRIAL: NCT02759744
Title: Pilot Study of Ultrasound Guided Focal Thermal Ablation of Prostate Cancer
Brief Title: Fusion Guided Focal Laser Ablation of Prostate Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 160098; 16-CC-0098
Record Dates: First submitted 2016-04-22; First posted 2016-05-03 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12-23

CONDITIONS: Prostate Cancer; Prostate Neoplasms
Keywords: Thermal Ablation; Localized Prostate Cancer; Medtronic-Visualase; Thermal Damage; PSA Levels
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): ultrasound image-guided focal ablation
  Interventions: Device: ultrasound image-guided ablation device

INTERVENTIONS:
Device: ultrasound image-guided ablation device — ultrasound image-guided focal ablation - may be either laser ablation or cryotherapy

SUMMARY:
Background:

Prostate cancer is the most common non-skin cancer in U.S. men. Treatments for early or less aggressive disease are limited. Researchers want to test a device that destroys cancerous tissue with laser energy. They want to see if using it with ultrasound is more comfortable than using it with magnetic resonance imaging (MRI).

Objectives:

To test a cooled laser applicator system to treat prostate cancer lesions. To see if ultrasound imaging is a practical and feasible treatment with laser ablation for focal prostate cancer treatment.

Eligibility:

Men at least 18 years old with prostate cancer seen on MRI that has not spread in the body.

Design:

Participants will be screened with standard cancer care tests. These can include physical exam, lab tests, and MRI. For the MRI, they lie in a machine that takes pictures. Participants will have a prostate biopsy. Needle samples will be taken from 12 places in the prostate. This will be guided by MRI and ultrasound, which is obtained through a coil in the rectum.

Participants will stay at the clinic for 1 2 days. A cooling catheter (plastic tube) will be put in the bladder. Ultrasound will guide the laser applicator directly to the tumor.

The cooling catheter will be removed. A different catheter will be put in the urethra to keep the bladder emptied.

The next day, participants will have a physical exam and a PSA blood test.

Participants will have 6 follow-up visits over 3 years. At each visit, they will have a physical exam and lab tests. At some visits, they will also have an MRI or other scans and a prostate biopsy.

DETAILED DESCRIPTION:
Background:

* Pilot study to evaluate the feasibility of real time ultrasound imaging to guide focal thermal ablation of low to intermediate risk focal prostate tumors.
* Prostate cancer is relatively slow growing, with doubling times for local tumors estimated at 2 to 4 years.
* Recent patient series suggest that 20% to 30% of men undergoing radical prostatectomy have pathologic features in the radical prostatectomy specimen consistent with an insignificant or "indolent" cancer that poses little threat to life or health.
* An NIH/NCI protocol #11-C-0158 titled MR Image guided focal laser ablation therapy of prostate cancer has treated 15 patients without major complication over the past 5 years. Out of 15 patients, 3 have had evidence of disease recurrence (data from this study was published in Diagnostic and Interventional Radiology). This data are being prepared for publication (verbal communication with Peter Pinto, MD, principal investigator); however, it requires a very long and resource-intensive MRI imaging, which may be a barrier to broad translation to the community setting. Specialized custom and expensive MRI-compatible equipment is also required. Focal laser ablation for prostate cancer using the Tranberg CLS Thermal Therapy System and laser are FDA cleared.
* Focal thermal ablation such as laser ablation or cryosurgery are standard of care therapies for prostate cancer, with cancer control comparable to that of external beam radiotherapy and brachytherapy.
* NIH / NCI clinical trials have performed MRI + ultrasound (US) fusion biopsy in nearly 3000 patients, > 40,000 biopsies over the past 18 years.
* We propose to perform ultrasound (US) guided focal thermal ablation with fusion visualization and co-display of pre-acquired MRI during the treatment of patients.

Objectives:

-To determine the feasibility of treating biopsy-confirmed, US-targetable and/or MR-visible, low to intermediate risk prostate tumor(s) using ultrasound (US) image-guided focal interstitial thermal ablation.

Eligibility:

* Patients must have organ confined, biopsy-confirmed, low or intermediate risk prostate cancer that is either US-targetable or MR visible, or both.
* Men >= 18 years of age.

Design:

* Pilot study, testing feasibility of ultrasound-guided thermal ablation of focal prostate cancer.
* A total of 30 patients will be enrolled to yield 20 evaluable patients

ELIGIBILITY:
* INCLUSION CRITERIA:
* Enrollment open only to current NIH patients enrolled in 16-C-0010.
* Patients

Patients must have clinically localized, non-aggressive, favorable or unfavorable, low to intermediate risk prostate cancer as defined per current NCCN guidelines (i.e, including review and determination of pathology and tumor characteristics, Gleason Score, PSA levels, and other assessments as clinically appropriate).Organ confined clinical prostate cancer that is US-targetable and/ or visualized on MRI or by a semi-automated software tool

* Prostate cancer diagnosed by transrectal or transperineal US-guided standard 12 core needle biopsy, MR image-guided needle biopsy, or MR/US fusion-guided needle biopsies or biopsies performed under semi-automated tools.
* Targeted tumors must be considered a safe distance (>= 8 mm) from the urethra, rectal wall, bladder wall or neurovascular bundle by the Principal Investigator.
* Must have had a prostate MRI performed at the NIH within 12 months prior to enrollment.
* Must have had a prostate biopsy performed at NIH within 12 months (+2 months) prior to enrollment.
* Men >18 years of age.
* ECOG performance status <=2.
* Patients must have adequate organ and marrow function as defined below:

  * leukocytes: >=3,000/mcL
  * absolute neutrophil count: >=1,500/mcL
  * platelets: >=75,000/mcL
  * creatinine: within normal institutional limits

OR

--creatinine clearance: >=60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

* Preoperative clearance by NIH Department of Anesthesia and Surgical Services
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Subject understands that this is an experimental protocol and that there are available standard treatment options. These options would include but not be limited to: active surveillance, external beam radiation and brachytherapy, androgen deprivation therapy, or prostatectomy.

EXCLUSION CRITERIA:

* Patient unable to commit to follow-up
* Acute urinary tract infection
* Patients with uncontrolled coagulopathies
* Altered mental status preventing consent or answering questions during conduct of the trial will be excluded for safety purposes
* A serious acute or chronic illness that is determined by the PI to place the patient at unreasonable risk for anesthesia and the procedure.
* Inability to undergo a contrast enhanced MRI per American College of Radiology and the Clinical Center, Department of Radiology guidelines.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the Principal Investigator, would limit compliance with study requirements.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of treating biopsy-confirmed and MR-visible, low-grade prostate tumor(s) using ultrasound (US) image-guided focal interstitial thermal ablation | duration of protocol
  Assessment of thermal damage outside of intended treatment areas as measured by post contrast MRI, and the frequency of other adverse events and complications.

SECONDARY OUTCOMES:
To determine changes in imaging and biopsy characteristics after thermal ablation of prostate cancer. | 3 years after treatment completed
To analyze circulating tumor markers and functional markers in individuals with prostate cancer after receiving treatment over time | 2 weeks after the ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-CC-0098.html